CLINICAL TRIAL: NCT01443819
Title: Randomized, Prospective Study of Lumbar Transforaminal Epidural Corticosteroid Injection(s) Versus Defined Physical Therapy for the Treatment of Subacute Lumbar Radicular Pain Due to Disc Protrusion
Brief Title: Lumbar Transforaminal Epidural Corticosteroid Injection(s) Versus Defined Physical Therapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment problem
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Matthew W Smuck, Principal Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SU-09232011-8446
Record Dates: First submitted 2011-09-26; First posted 2011-09-30 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Lumbar Radiculopathy
Keywords: Radiculopathy; Transforaminal; Disc Protrusion
MeSH Terms: conditions — Radiculopathy; Intervertebral Disc Displacement | interventions — Physical Therapy Modalities; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lumbar Transforaminal Epidural Corticosteroid Injection (Other)
  Interventions: Other: Lumbar Transforaminal Epidural Corticosteroid Injection
- Physical Therapy (Other)
  Interventions: Other: Physical Therapy
- Cohort observational (Other)
  Interventions: Other: Observation

INTERVENTIONS:
Other: Lumbar Transforaminal Epidural Corticosteroid Injection — Injection: Anesthetic/corticosteroid (per randomization); repeat 1-3 times if clinically indicated.
  The following drugs will be used for this procedure: 80mg Depo-Medrol and 1% lidocaine. These drugs used for the epidural injections are local anesthetic numbing medicines and cortisone/steroid anti-inflammatory medicines.
  Arms: Lumbar Transforaminal Epidural Corticosteroid Injection
Other: Physical Therapy — Physical therapy carried out per protocol; 2-3 times per week for a total of 12 treatment sessions (excluding initial evaluation, including exit evaluation, minimum attendance 8/12) to be completed by 6 weeks from initiation of care (within study).
  Please note: There will be another PT evaluation at the end of 6 weeks.
  Arms: Physical Therapy
Other: Observation — If subject declines then inquire about enrolment in the observational cohort. Participants in this group (Cohort) will chose their treatment (per-protocol physical therapy, injections, or both) after consulting with their physicians.
  Arms: Cohort observational

SUMMARY:
The purpose of this research study is to look at two of the common forms of treatment for this condition: physical therapy and epidural steroid injection. The investigators are attempting to evaluate whether or not physical therapy alone, or epidural steroid injections alone, are effective in treating this condition. The investigators will also try to determine whether or not one of these treatments is better than the other for the treatment of herniated discs with nerve injury (radiculopathy).

DETAILED DESCRIPTION:
1. Potential research participants identified from clinic population.

   * 40 subjects will be enrolled in each group (TFESI and PT). An additional 40 subjects will be enrolled into the concurrent observational cohort.
   * Appropriate study subjects will be identified upon initiation of care (MD evaluation and/or physical therapy). They will have pain of less than or equal to three months duration, within the current pain episode. This may be the initial pain episode or the onset of a most recent episode of pain, preceded by at least a six month pain free interval. They will have focal disc protrusion with correlating radicular symptoms and possible radicular/neurological deficits. These radicular symptoms/signs are defined as pain or paresthesias below the knee, pain reproduction with straight-leg-raising and/or extension or quadrant maneuvers, and radicular pattern sensory, reflex or strength changes. These symptoms will be consistent with the level of nerve root impingement. Only subjects with radiculopathy primarily at L5 and/or S1, due to pathology at L4-5 and/or L5-S1 disc levels will be included. Those with canal and foraminal compromise due to disc protrusion at L4-5 with L5 > L4 signs and symptoms WILL be included. Those with predominantly degenerative stenosis, degenerative spondylolisthesis, or spondylolysis will be excluded.

   Subjects also need to have an eleven point Likert pain scale score greater than or equal to four. They will not have a history of prior epidural steroid injections within the prior year or prior lumbar surgery.
2. Initial evaluation and study eligibility determination.
3. Presentation of study to patient and informed consent obtained
4. Baseline pain and outcome measures evaluation (VAS, SF-36, ODI, GPC, PSAQ, physical exam, work history, analgesic use log, and ancillary treatment log, lost productivity).

   -Upon entry to the study, baseline measurements of the patient's pain and function will be established. The primary outcome measure for this study will be reduction in pain as measured by a three day average Visual Analog Scale (VAS). Secondary measures will include: Oswestry Disability Index (ODI), SF-36, a seven point Global Perception of Change (GPC), a three question Patient Specific Activity questionnaire (PSAQ) (each patient will list 3 cardinal activities of daily living that are restricted or rendered impossible because of their pain and will score each item), and utilization of analgesic, outside medical care, and surgical options, as well as physician physical exam test parameters and lost productivity.
5. Randomization to TFESI or PT group, if subject declines then inquire about enrolment in the observational cohort. Participants in this group (Cohort) will chose their treatment (per-protocol physical therapy, injections, or both) after consulting with their physicians.
6. Injection: Anesthetic/corticosteroid (per randomization); repeat 1-3 times if clinically indicated.

   The following drugs will be used for this procedure: 80mg Depo-Medrol and 1% lidocaine.

   These drugs used for the epidural injections are local anesthetic numbing medicines and cortisone/steroid anti-inflammatory medicines.
7. Physical therapy carried out per protocol; 2-3 times per week for a total of 12 treatment sessions (excluding initial evaluation, including exit evaluation, minimum attendance 8/12) to be completed by 6 weeks from initiation of care (within study).

   Please note: There will be another PT evaluation at the end of 6 weeks.
8. MD visit at intake evaluation, 4 weeks, 12 weeks,6 months, 12 months (additional phone contact or prn follow up will be logged as additional care)
9. Pain and functional evaluations at: baseline, 4 weeks, 12 weeks, 6 months, 12 months (VAS, SF-36, ODI, GPC, PSAQ, work history, analgesic use log, lost productivity and ancillary treatment log).

   * At the 4 week follow-up, subjects who are not satisfied with treatment will be provided the option to cross-over to the alternate treatment group.

Participants in the control group will chose their treatment (per-protocol physical therapy, injections, or both) after consulting with their physicians.

All of the procedures for this protocol are standard of care.

We will be asking participants if they are willing to be contacted regarding future research studies that may be of interest to them.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion highlights: L4-5 or L5-S1 HNP with leg>back pain; duration < 12 weeks.

1. Low back pain episode less than or equal to 12 weeks in duration, within the current pain episode. This may be the initial pain episode or the onset of a most recent episode of pain, preceded by at least a six month pain free interval.
2. Visual analog score (VAS) or screening Likert pain scale score three day average and present pain of at least four/ten at baseline.
3. Age 18 to 64.
4. Subjects will have focal disc herniation with unilateral radicular/neurological deficits or correlating radicular symptoms. These radicular symptoms/signs are defined as pain or paresthesias below the knee, pain reproduction with straight-leg-raising and/or extension or quadrant maneuvers, and radicular pattern sensory, reflex or strength changes. These symptoms will be consistent with their level of nerve root impingement and will primarily involve the L5 and/or S1 roots.
5. Those with canal and foraminal compromise due to disc herniation at L4-5 with L5 > L4 signs and symptoms WILL be included.

Exclusion Criteria:

1. Litigation.
2. Workers compensation.
3. Those receiving remuneration for their pain, e.g. disability.
4. Back pain greater than leg pain.
5. Scoliosis of > 15 degrees
6. Those unable to read English and complete the assessment instruments.
7. Spondylolysis, with or without spondylolithesis, degenerative spondylolithesis, or stenosis due primarily to degenerative bony or soft tissue changes.
8. Systemic inflammatory arthritis (e.g. rheumatoid, lupus).
9. Addictive behaviour, severe clinical depression, or psychotic features.
10. Significant lower extremity pathology that effects gait.
11. Sustained cervical or thoracic pain that is present at a level >4/10 on VAS.
12. Possible pregnancy or other reason that precludes the use of fluoroscopy.
13. Prior lumbar surgery
14. Prior epidural steroid injections for treatment of current episode or within the prior year
15. Bilateral radicular signs/symptoms (< 90% laterality of pain intensity or bilateral neurological signs)
16. No more than 4 PT sessions for current episode

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score | 12months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Smuck, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Spinal Diagnostics and Treatment Center, Daly City, California
  - Comprehensive Spine and Sport, Mill Valley, California
  - Stanford University Medicine Outpatient Center, Redwood City, California